CLINICAL TRIAL: NCT06449404
Title: 7.0T Magnetic Resonance Imaging Study of Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Director and Clinical Professor, Chinese PLA General Hospital
Other Study IDs: Parkinson's disease-ChinaPLAGH
Record Dates: First submitted 2022-03-14; First posted 2024-06-10 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Parkinson's Diseases; MRI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 7T-MRI scaning — 7T-MRI scaning

SUMMARY:
This clinical trial study is conducted to detect the imaging characteristics of the patients with Parkinson's diseases (PD) by 7-Tesla (7T) magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
In this study,we explored the imaging characteristics of PD. First, with the advantage of 7T, we detect the slight changes of PD with short diseases history compared with the healthy. Second, we investigate the different imaging characteristics in subtypes of PD, finding the effective neuroimaging biomarkers to distinguish different subtypes of PD. Finally, we take long time follow-up to evaluate the correlation between the imaging changes and clinical score alteration in PD.

ELIGIBILITY:
Inclusion Criteria:

* the patients with PD who was diagnosed by the experienced neurologist specializing in movement disorders

Exclusion Criteria:

* the patients with brain disorders such as cerebrovascular disease, brain tumors, epilepsy, other neurodegenerative disease;
* psychiatric disorders with impaired cognitive function;
* contraindications to MRI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
The change in motor symptoms in PD patients. | 5 year after the conduction of clinical trial
  The patient's clinical state was evaluated according to the Movement Disorder Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) and H-Y scale. The former scale total score ranges from 0 to 199, with higher scores indicating more severe symptoms in patients. H-Y scale categorizes PD into five stages with higher stages indicate more severe symptoms.
  Comparison will be performed from examinations for case-control study versus for baseline and 5-year follow-up timepoints.

SECONDARY OUTCOMES:
Functional connectivity alterations between individuals with different subtypes of PD and healthy subjects. | 5 year after the conduction of clinical trial
  The functional connectivity calculation is primarily based on the BOLD sequence, which is used to describe the degree of connectivity between different brain regions, reflecting the functional activity of the brain. A higher value indicates stronger connectivity and more active function.
Structural connectivity alterations between individuals with different subtypes of PD and healthy subjects. | 5 year after the conduction of clinical trial
  The structural metrics calculation is primarily based on the MP2RAGE and DTI sequence, which is used to describe cortical thickness, subcortical nuclei volume, as well as the connectivity of white matter connectivity, respectively. A higher value indicates larger thickness (volume) or stronger connectivity.
Clinical variables spectrum features linking to the motor symptoms and imaging spectrum features. | 5 year after the conduction of clinical trial
  Medical records and test data of patients, including demographic characteristics, motor scores, non-motor scores, common comorbidity, hematological analysis, coagulation function, lipids profile, blood biochemistry, were used to construct clinical variables spectrum features. The distribution characteristics of motor symptoms and imaging spectrum features were compared with the multi-dimensional matrix. Gene-imaging association analysis was also used to evaluate the imaging changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing, China, China

IPD SHARING:
Plan to Share IPD: Undecided